CLINICAL TRIAL: NCT03669198
Title: A Health Economic Evaluation of Using N-Terminal Pro Brain Natriuretic Peptide (NT-pro BNP) for Management of Acute Heart Failure in a Tertiary Referral Hospital in Jakarta, Indonesia
Brief Title: A Health Economic Evaluation of Using N-Terminal Pro Brain Natriuretic Peptide (NT-Pro BNP) in Acute Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Failure Biomarker Group (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HFBG
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Heart Failure
Keywords: Acute Heart Failure; Cost; NT-pro BNP
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NT-pro BNP group (Active Comparator): Subjects who be included in NT-pro BNP group examined NT-pro BNP in the ED to determine the baseline level and prior to discharge for determine the percent decline from baseline level. Patients in the NT-pro BNP group can be discharged if the NT-pro BNP level decreased ≥ 30% from baseline. If the target percent decline is not met, we will do intensification of therapy according to the algorithm
  Interventions: Diagnostic Test: NT-Pro BNP
- Control group (No Intervention): Patients in the control group were managed based on clinical judgment without use of NT-pro BNP testing. In the control group, the decision whether patient can be discharged or not was determined by cardiologist in charge of the patient based on clinical assessment.

INTERVENTIONS:
Diagnostic Test: NT-Pro BNP — . AHF patients who met inclusion and exclusion criteria were randomly assigned to 2 groups, NT-pro BNP group and control group. In the NT-pro BNP group, serial NT-pro BNP levels at admission and pre-discharge was measured, the latter with the target of decrease ≥ 30% NT-pro BNP level. Randomised patients were followed during treatment up to 90 days post-discharge to assess short-term outcomes and costs.
  Other Names: Natriuretic peptide
  Arms: NT-pro BNP group

SUMMARY:
Cardiac biomarkers have dramatically impacted the way HF patients are evaluated and managed. In fact, the role of biomarkers has developed to better differentiate HF against other diseases and, to timely initiate and influence more accurate diagnosis (rule out) and treatments, to predict the onset of future HF, to risk-stratify affected patients, and to serve as a tool to guide intensity of therapy. NT-proBNP has become validated biomarkers with highest guideline recommendation (class I) and independent predictors for re-hospitalization and mortality in HF patients. However, many Indonesian cardiologists do not use of those biomarkers, mostly due to limited available cardiac biomarkers for the cost effective heart failure management. We evaluate 2 alternative treatments which one that more cost-effective between biomarker's guided therapy and without biomarker.

DETAILED DESCRIPTION:
With growing demands on limited health care budgets, optimal resource allocation in HF patients is essential. Although NT pro BNP is proposed to be effective for the evaluation and management patients with heart failure, no data exist about cost-effectiveness analysis that are based on practice patterns endorsed by universal coverage systems in Indonesia (Jaminan Kesehatan Nasional). Because NT-proBNP therapy guidance in HF is believed to create additional costs, it is not yet broadly applicable. Its why we need to elaborate this issue.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years
* The primary diagnosis at the Emergency Department (ED) is acute decompensated heart failure (ADHF)
* Using the national health insurance
* Willing to be followed for 3 months
* Willing to sign informed consent.

Exclusion Criteria:

* Severe life-threatening comorbidities with a life expectancy of <2 years
* Acute heart failure other than ADHF such as acute pulmonary edema, acute heart failure in the setting of acute coronary syndrome, cardiogenic shock, right heart failure, and hypertensive heart failure
* ADHF accompanied by sepsis, liver disease, lung disease with severe radiological findings, mechanical complications of acute myocardial infarction, aortic dissection, congenital heart disease, idiopathic pulmonary hypertension, lung emboli, severe respiratory failure, and severe burns
* Patients admitted to ICVCU (Intensive Cardiovascular Care Unit)
* Patients did not take medication regularly and controls routinely.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 3 months after discharge
  Percentage of patients who are death post discharge (%)
Rehospitalization rate | 3 months after discharge
  Percentage of patients who readmit and are hospitalized because of heart failure (%)
Emergency department visit | 3 months after discharge
  Percentage of patients who readmit and are not hospitalized because of heart failure (%)

SECONDARY OUTCOMES:
Cost | Admission to hospital until 3 months after discharge
  Total cost include cost of hospitalization, cost of rehospitalization and cost of emergency department visit (Rupiah)

CONTACTS AND LOCATIONS:
Overall Officials: Prima Almazini, MD, Principal Investigator — Heart Failure Biomarker Group
Locations (1):
- Heart Failure Biomarker Group, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
IPD are not to be shared with other researchers